CLINICAL TRIAL: NCT05688592
Title: A Prospective Multicenter Study to Determine the Usefulness of Systematic 18-FDG-PET-TC for the Management of Invasive Fungal Infection (PETIFI Project)
Brief Title: Usefulness of PET-CT for Invasive Fungal Infection
Acronym: PETIFI
Status: Recruiting | Type: Observational
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Ana Fernandez Cruz, MD, PhD, Puerta de Hierro University Hospital
Other Study IDs: GLD22/00032
Record Dates: First submitted 2022-12-20; First posted 2023-01-18 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Invasive Fungal Infections
Keywords: invasive fungal infection; PET-CT; management; staging; monitoring response
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Controlled Before-After Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PET-CT — This is a before-and-after study (not a clinical trial)
  * in the case of fungemia, 2 weeks after the initial staging 18F-FDG PET-CT.
  * in the case of focal IFIs, 2-4 and 12 weeks after the initial staging 18F-FDG PET-CT
  Other Names: Before-and-after study

SUMMARY:
The goal of this national multicenter prospective cohort study is to learn about the added value of 18F-FDG (18F-2-fluoro-2-deoxy-D-glucose) PET-CT in invasive fungal disease management. The main questions it aims to answer are:

1. Does the use of 18F-FDG PET-CT allow a better characterization of invasive fungal infection (IFI) (performance) compared to the exclusive use of conventional radiological studies in terms of extension/staging and monitoring of response/follow-up ?
2. Does the systematic and protocolized use of 18F-FDG PET-CT in IFI allow a better management of patients with IFI and increase the prognostic value of the initial evaluation? Participants will undergo systematically a 18F-FDG PET-CT as part of the work-up of their invasive fungal disease. Researchers will compare the performance of 18F-FDG PET-CT with standard management without 18F-FDG PET-CT to see if adds value (diagnostic, prognostic, and changes in management).

DETAILED DESCRIPTION:
Design: National multicenter prospective cohort study . Participating centers: 14 Spanish tertiary hospitals (see work plan)

For inclusion in the study, two types of IFIs will be considered:

* IFI in the form of fungemia: detection of fungal growth in blood cultures.
* Focal IFI with tissue invasion: patients with a diagnosis of proven or probable IFI according to the corresponding criteria depending on the type of patient (Hematology and other immunocompromised: European Organization for Research and Treatment of Cancer (EORTC)/Mycoses Study Group Education and Research Consortium (MS GERC) consensus definitions; solid organ transplantation: 2010 International Society for Heart and Lung Transplantation (ISHLT) consensus statements for the definitions of infections in cardiothoracic transplant recipients; ICU/Chronic obstructive pulmonary disease: Bulpa criteria; COVID-19 (Coronavirus disease-2019): ECMM (European Confederation of Medical Mycology)/ISHAM.

Sample size:

Based on the literature, we assume that 18F-FDG PET-CT will detect lesions not previously visualized in approximately 50% of patients (7). We anticipate that the findings in 50% of these patients will cause the management of IFI to change, which corresponds to 25% of the total number of patients. To achieve a 6% accuracy in estimating a proportion using a bilateral 95% Normal asymptotic confidence interval, assuming that the proportion is 25%, it will be necessary to include 201 patients in the study. Assuming 10% of abandonments, or loss of information, it would be necessary to recruit 224 patients.

Period of inclusion of patients in the study: 2 years Patient Recruitment Upon suspicion of IFI, the attending physician will verify that the patient meets all the inclusion criteria and none of the exclusion criteria and will contact Nuclear Medicine to schedule the performance of 18F-FDG PET-CT according to the deadlines established in the study protocol.

Intervention

In addition to the usual management (detailed below) 18F-FDG PET-TC will be performed to evaluate:

* staging at diagnosis: in the first week after diagnosis (preferably in the first 48 hours of starting antifungal treatment).
* response monitoring/follow-up: will be carried out on the same equipment as the initial 18F-FDG (18F-2-fluoro-2-deoxy-D-glucose).

PET-TC

* in the case of fungemia, 2 weeks after the initial staging 18F-FDG PET-CT.
* in the case of focal IFIs, 2-4 and 12 weeks after the initial staging 18F-FDG PET-CT.

Data collection and analysis The information shall be collected prospectively by means of a data collection notebook (eDCN) and stored in an anonymized form in a common database specially designed for the study The data will be obtained from the patient's medical history of the different participating centers. From the database, they will be downloaded to the statistical program for analysis, which will be carried out with the support of the Biostatistics Unit of Instituto de Investigación Puerta de Hierro-Segovia did Arana (IDIPHISA).

Demographic, clinical variables, and results of conventional diagnostic tests including blood count, biochemistry, cultures according to presentation, biomarkers such as galactomannan or D-glucan, and imaging tests (x-rays, CT, MRI or echocardiogram) performed according to clinical indication (standard of care, SOC) and following the guidelines will be collected. Specifically, anatomy-based imaging tests will be performed according to the protocols of each department, and will be interpreted by certified specialists (radiologists, echocardiographists, etc ... as appropriate) as part of routine care.

Analysis of 18F-FDG PET-CT images:

In order to standardize the interpretation of the images in the different participating centers, a one-day training session will be held before the start of the study with the participation of all the Nuclear Medicine doctors involved in the project.

The 18F-FDG PET-CT will be reviewed by the specialist of the patient's center who will be blind to the result of the tests performed according to standard of care (SOC). Additionally, the images will be included in the database, for evaluation by a second specialist in Nuclear Medicine from the coordinating center, blind for the initial interpretation of the 18F-FDG PET-TC.

This second evaluation will favor the standardization of the interpretation, however, for reasons of time and opportunity, clinical decisions will be made based on the interpretation of the local Nuclear Medicine team.

Pre-PET (Pre-18F-FDG PET-TC ) evaluation:

* Staging

  * In this phase, IFIs will be classified into localized or disseminated disease (involvement of more than one non-contiguous organ; in the case of fungemia, detection of septic metastases), and the number of lesions and organs affected will be specified.
  * Prior to the completion of the initial 18F-FDG PET-CT, the attending physician will establish a staging and management plan of the IFI based on the data known at that time, through a standardized questionnaire: need for diagnostic techniques, source control (including surgical treatment), selected drug (penetration into involved areas, need for combined treatment), expected duration of treatment.
* Response monitoring (follow-up):

  * The relevant clinical, analytical, microbiological and imaging tests performed at the time of the 18F-FDG PET-CT follow-up will be collected. Additional tests will be performed according to. clinical indication (SOC).
  * An evaluation of the response to treatment and management plan of the IFI will be established prior to the performance of the 18F-FDG PET-TC (pre-PET) (including prevision to discontinue or maintain antifungal).

Post-PET (Post-18F-FDG PET-TC ) evaluation

* Staging

  * Based on the findings of the 18F-FDG PET-CT, IFIs will be classified again in localized or disseminated disease, and the number of lesions and organs involved will be specified.
  * The contributions of the 18F-FDG PET-TC to the data that were known prior to its realization will be specifically collected, as well as the specific data of the 18F-FDG PET-TC (SUV max, ....).
* Response monitoring -After the PET, a re-evaluation of the response to the treatment will be established based on the PET findings and, in the first 48 hours after the performance and evaluation of the initial 18F-FDG PET-CT, the same responsible physician will reevaluate the management plan based on the findings of the 18F-FDG PET-CT establishing the modifications it deems necessary. Clinical decisions will be made based on the interpretation of the local Nuclear Medicine team.

The patient's outcome will be evaluated at 100 days and 6 months (completion of treatment, continuation of chemotherapy or performance of stem cell transplantation (SCT), recurrence, survival).

Study variables (performance, clinical impact and evolution, according to the objectives)

1. Performance variables: percentage of patients with IFI in whom 18F-FDG PET-CT has improved patient assessment compared to standard management in:

   1. Initial staging of infection: change in staging (localized/disseminated); change in number of organs involved or number of fungal lesions detected. (number of lesions discordant between pre-PET and post-PET).
   2. Response to treatment: change in the assessment of the IFI response (clinical response, anatomical response, metabolic response)
2. Clinical impact variables: added value (patients benefiting from PET)

   1. 18F-FDG PET-CT will be considered to have added value over SOC when lesions are detected outside the region assessed by other imaging tests (7), clinically hidden lesions, dissemination, PET "reclassifies" a radiological finding (8) or leads to the performance of a new targeted diagnostic test.
   2. When the metabolic information provided by the 18F-FDG PET-CT allows clinical decisions about the patient to be made, either to discontinue, prolong or change the anti fungal treatment (modification of the type of treatment, modification of the drug used, modification of the duration of treatment) or leads to surgical treatment, it will be considered to be modification of the treatment and has added value.
   3. Added value shall be considered when baseline metabolic parameters allow predicting metabolic response to anti fungal therapy.

ELIGIBILITY:
Inclusion criteria:

* 18-year-old adult patients
* who are admitted with a diagnosis of invasive fungal infection
* who able to undergo a one 18F-FDG PET-CT
* who give their informed consent.

Exclusion criteria:

* concomitant active bacterial infection likely to produce uptake in organs and tissues
* recent surgery in the area of the IFI (in the previous 3 months)
* other medical conditions that interfere with the development of the study ( e.g., inability to tolerate the performance of the test during the required time, pregnancy)
* terminal situation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted with a diagnosis of invasive fungal infection, both fungemia or focal fungal infection
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Duration of antifungal treatment | 6 months
  Length of anti fungal therapy
Survival | 6 months
  Alive at the last visit

SECONDARY OUTCOMES:
Resumption of chemotherapy or performance of stem cell transplantation | 6 months
  The infection recedes enough to allow the receipt of chemotherapy
Recurrence of invasive fungal infection | 6 months
  New episode of fungal infection caused by the same pathogen

CONTACTS AND LOCATIONS:
Overall Officials: Ana Fernández Cruz, MDPhD, Principal Investigator — Hospital Puerta de Hierro-Majadahonda
Locations (14):
- Spain (14):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madriid
  - Hospital de Bellvitge, Barcelona
  - Hospital Universitario Clinic, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Infanta Leonor Hospital, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Unversitario Ramón y Cajal, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Messeguer, Murcia
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Unversitario de Salamanca, Salamanca
  - Hospital Universitario Virgenn de la Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication
Access Criteria: The Individual Patient Data underlying results in a publication will be shared

REFERENCES:
- [Derived] Gutierrez A, Rodriguez B, Velasquez K, Gutierrez I, Garcia S, Munez E, Calderon-Parra J, Callejas-Diaz A, Ramos-Martinez A, Fernandez-Cruz A. Determining the usefulness of systematic 18F-FDG PET/CT for the management of invasive fungal infection (PETIFI project): a prospective national multicentre cohort study protocol. BMJ Open. 2023 Jun 23;13(6):e074240. doi: 10.1136/bmjopen-2023-074240. PMID 37355275